CLINICAL TRIAL: NCT05912569
Title: Feasibility Study on Delayed Selective Sentinel Node Biopsy for Patients Undergoing Mastectomy for Ductal Carcinoma in Situ
Brief Title: Delayed Selective Sentinel Node Biopsy for Patients Undergoing Mastectomy for DCIS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Hyeong-Gon Moon, Professor, Seoul National University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2212-088-1386
Record Dates: First submitted 2023-06-12; First posted 2023-06-22 (Actual); Last update posted 2025-01-31 (Actual); Status verified 2025-01

CONDITIONS: DCIS
MeSH Terms: conditions — Carcinoma, Intraductal, Noninfiltrating

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Delay sentinel node biopsy (Experimental): sinlge arm
  Interventions: Procedure: Delay sentinel node biopsy

INTERVENTIONS:
Procedure: Delay sentinel node biopsy — In the case of a patient undergoing breast-conserving surgery for intraductal carcinoma, the sentinel lymph node is not excised during the primary surgery but only marked for identification. I

SUMMARY:
In the case of a patient undergoing total mastectomy for intraductal carcinoma (DCIS), the sentinel lymph node is not excised during the primary surgery but only marked for identification. If the final histological examination confirms invasive cancer, delayed surgery is performed to remove the sentinel lymph node that was marked during the initial surgery.

primary endpoint : The success rate of identifying the sentinel lymph node that was marked during the primary surgery in cases where the final histological examination confirms invasive cancer is evaluated.

addendum) The previously documented Breast-Conserving Surgery has been corrected to reflect the accurate procedure of Total Mastectomy.

DETAILED DESCRIPTION:
Primary surgery:

Patients diagnosed with intraductal carcinoma through histological examination and scheduled for axillary lymph node dissection are included.

Prior to the surgery, blue dye and/or radioisotope injection are used to identify the sentinel lymph node, similar to the current practice.

total mastectomy surgery is performed. After identifying the sentinel lymph node in the axillary region, its location is marked using a titanium clip (size 2-4mm) or sutures (Maxon 3-0, a slow monofilament absorbable suture).

The number of marked sentinel lymph nodes is recorded for documentation.

Confirmation of pathological examination results:

If the final surgical specimen confirms invasive carcinoma (size > 1mm) through pathological examination, sentinel lymph node surgery is performed.

addendum)

1. Suture Specification The surgical procedure will utilize Maxon 3-0, a slow monofilament absorbable suture for optimal tissue approximation and healing.
2. Management of Microinvasive Cancer For cases where the tumor size is 1 mm or smaller (microinvasive cancer), the decision to proceed with reoperation will be made at the discretion of the treating physician based on clinical judgment.

Secondary surgery:

Prior to the surgery, an axillary view x-ray is taken to verify the location and number of the clips.

Blue dye and/or radioisotope injection is administered near the axillary incision site.

Accessing the axillary region involves identifying the marked areas using clips or sutures and detecting sentinel lymph nodes for biopsy.

The number of removed clips/sutures and the number of sentinel lymph nodes identified are documented for record keeping.

addendum) Axillary X-ray and Sentinel Node Mapping Axillary x-ray and the use of blue dye or radioisotope injection for sentinel lymph node mapping are not mandatory and may be utilized at the physician's discretion.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 20 to 75 years old.
* Patients diagnosed with DCIS through histological examination.
* Patients undergoing mastectomy

Exclusion Criteria:

* In cases where the histopathological findings of the tissue examination indicate suspicious invasive lesions.
* In cases where imaging tests or physical examinations suggest possible lymph node metastasis.
* In patients who have previously undergone axillary lymph node surgery on the same side as the current procedure.
* Pregnant patients.

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2023-06-13 (Actual); Primary Completion 2025-04-28 (Estimated); Study Completion 2025-04-28 (Estimated)

PRIMARY OUTCOMES:
success rate | 2 weeks later
  The success rate of identifying the sentinel lymph node that was marked during the primary surgery in cases where the final histological examination confirms invasive cancer is evaluated.

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Yes